CLINICAL TRIAL: NCT01142622
Title: Do Peritoneal Nebulization of Ropivacaine Reduce the Use of Morphine After Short Gynecologic Laparoscopic Surgery?
Brief Title: Intraperitoneal Ropivacaine Nebulization for Pain Control After Gynecologic Laparoscopic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: San Gerardo Hospital (Other)
Collaborators: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Pablo Mauricio Ingelmo M.D., Consultant Anesthesiologyst, San Gerardo Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR HSG 02 2010 Ovarian Cyst
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Ovarian Cysts
Keywords: Ovarian Cysts; Nebulization; Ropivacaine
MeSH Terms: conditions — Ovarian Cysts | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine nebulization (Experimental): Preoperative nebulization of 150 mg of Ropivacaine in the peritoneal cavity
  Interventions: Drug: Ropivacaine nebulization
- Ropivacaine instillation (Active Comparator): Preoperative instillation of 150 mg of Ropivacaine in the peritoneal cavity before surgery
  Interventions: Drug: Ropivacaine instillation

INTERVENTIONS:
Drug: Ropivacaine nebulization — Preoperative nebulization of 150 mg of Ropivacaine in the peritoneal cavity.
  Other Names: Ropivacaine; Nebulization
  Arms: Ropivacaine nebulization
Drug: Ropivacaine instillation — Preoperative instillation of 150 mg of Ropivacaine in the peritoneal cavity.
  Other Names: Ropivacaine; Instillation
  Arms: Ropivacaine instillation

SUMMARY:
The purpose of this study is to assess if intraperitoneal nebulization of Ropivacaine 150 mg may prevent the use of morphine during the first day after laparoscopic ovarian cyst surgery.

DETAILED DESCRIPTION:
In a recent study the investigators found that nebulization of Ropivacaine 30 mg before or after gynaecologic laparoscopic surgery significantly reduces postoperative pain and postoperative morphine consumption.

Ropivacaine was effectively administered with non-heating nebulizers (AeronebPro®).

However, almost all patients still use morphine after surgery.

The investigators hypothesize that intraperitoneal nebulization of Ropivacaine 150 mg may prevent the use of morphine after the laparoscopic ovarian cyst surgery.

ELIGIBILITY:
Inclusion Criteria:

* Females 18-65 years old
* ASA Score I-III
* Scheduled for ovarian cyst laparoscopic surgery
* Free from pain in preoperative period
* Not using analgesic drugs before surgery
* Without cognitive impairment or mental retardation
* Written informed consent

Exclusion Criteria:

* Emergency/urgency surgery
* Postoperative admission in an intensive care unit
* Cognitive impairment or mental retardation
* Progressive degenerative diseases of the CNS
* Seizures or chronic therapy with antiepileptic drugs
* Severe hepatic or renal impairment
* Pregnancy or lactation
* Allergy to one of the specific drugs under study
* Acute infection or inflammatory chronic disease
* Alcohol or drug addiction

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Morphine consumption (mg) | Up to 24 hours
  The total dose of morphine at every evaluation after awakening will be quantified using the PACU clinical chart and/or PCA infusers memory display.

SECONDARY OUTCOMES:
Postoperative Pain | Up to 24 hours
  Postoperative pain will be assessed by numeric ranking scale (NRS 0 to 10 points) at rest (static NRS) and after deep inspiration or cough (dynamic NRS). Pain after surgery will be differentiated as abdominal, wall pain, port wound pain, back pain and shoulder pain. The proportion of patients with adequate pain control after surgery (dynamic NRS < 3) will also be assessed.
Time of unassisted walking | Up to 24 hours
  Unassisted walking time is defined as the time in hours between PACU discharge and when the patient is able to walk out of his room and back to bed without any assistance.
Hospital morbidity | Up to 24 hours
  All complications or adverse effects associated or possibly associated with the interventions under study, surgery or anesthesia, will be quantified using the anesthesia charts, surgical charts and surgical database.
Hospital stay | Up to 24 hours
  We define hospital stay as the time in hours elapsed between surgery and hospital discharge. We evaluate the hospital stay with the post-anesthetic discharge scoring system (Modified-PADSS).
Quality of life after surgery | Four weeks after surgery
  Quality of life will be assessed using the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pablo M Ingelmo, MD, Principal Investigator — San Gerardo Hospital, Monza. Italy
Locations (1):
- San Gerardo Hospital, Monza, MB, Italy

REFERENCES:
- [Background] Greib N, Schlotterbeck H, Dow WA, Joshi GP, Geny B, Diemunsch PA. An evaluation of gas humidifying devices as a means of intraperitoneal local anesthetic administration for laparoscopic surgery. Anesth Analg. 2008 Aug;107(2):549-51. doi: 10.1213/ane.0b013e318176fa1c. PMID 18633034
- [Background] Alkhamesi NA, Peck DH, Lomax D, Darzi AW. Intraperitoneal aerosolization of bupivacaine reduces postoperative pain in laparoscopic surgery: a randomized prospective controlled double-blinded clinical trial. Surg Endosc. 2007 Apr;21(4):602-6. doi: 10.1007/s00464-006-9087-6. Epub 2006 Dec 16. PMID 17180268
- [Background] Schlotterbeck H, Schaeffer R, Dow WA, Diemunsch P. Cold nebulization used to prevent heat loss during laparoscopic surgery: an experimental study in pigs. Surg Endosc. 2008 Dec;22(12):2616-20. doi: 10.1007/s00464-008-9841-z. Epub 2008 Mar 18. PMID 18347861